CLINICAL TRIAL: NCT02509728
Title: Nahrungsergänzung Mit Cholin- Und Docosahexaensäure Bei Sehr Unreifen Frühgeborenen
Brief Title: Metabolic Effects of Choline and Docosahexaenoic Acid Supplementation in Preterm Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Choline and DHA for Preemies 2
Record Dates: First submitted 2015-07-22; First posted 2015-07-28 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Infant, Premature
Keywords: choline; docosahexaenoic acid
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- standard nutrition (Active Comparator): standard nutrition
  Interventions: Dietary Supplement: standard nutrition
- choline supplementation (Experimental): in addition to standard nutrition: enteral supplementation with 30mg/kg choline chloride for 10 days
  Interventions: Dietary Supplement: choline supplementation; Dietary Supplement: standard nutrition
- DHA supplementation (Experimental): in addition to standard nutrition: enteral supplementation with 60mg/kg DHA for 10 days
  Interventions: Dietary Supplement: DHA supplementation; Dietary Supplement: standard nutrition
- choline and DHA supplementation (Experimental): in addition to standard nutrition: enteral supplementation with 30mg/kg choline chloride and 60mg/kg of DHA for 10 days
  Interventions: Dietary Supplement: choline supplementation; Dietary Supplement: DHA supplementation; Dietary Supplement: standard nutrition

INTERVENTIONS:
Dietary Supplement: choline supplementation — in addition to standard nutrition: enteral supplementation with 30mg/kg choline chloride for 10 days
  Arms: choline and DHA supplementation; choline supplementation
Dietary Supplement: DHA supplementation — in addition to standard nutrition: enteral supplementation with 60mg/kg DHA for 10 days
  Arms: DHA supplementation; choline and DHA supplementation
Dietary Supplement: standard nutrition — standard nutrition

SUMMARY:
To explore the effects of enteral choline and DHA supplementation on plasma choline and DHA-PC concentrations and metabolism, this randomized controlled study will assign 40 preterm infants to 1 of 4 groups: standard care, choline supplementation, DHA supplementation, and choline and DHA supplementation.

After 7 days of supplementation, a single dose of stable isotope labelled choline will be administered and the kinetics of newly synthesized DHA-PC determined to assess plasma levels, uptake and distribution of choline and DHA.

This study is designed to inform larger studies evaluating this approach of enteral co-application of choline and DHA on clinical important outcomes.

DETAILED DESCRIPTION:
In utero, there is a constant high supply of choline to the fetus. Preterm delivery disrupts this maternal-fetal choline-transfer. We have shown that choline plasma levels rapidly half after preterm delivery. We also demonstrated that plasma DHA-PC rapidly falls after preterm delivery. DHA supplementation has been evaluated and found safe, however the clinical benefits have been smaller than expected. We speculate that choline deficiency may have contributed to the smaller than expected benefit of DHA supplementation in the past.

This study verifies the hypothesis that concomitant supply of choline and DHA will improve DHA-PC availability and turn-over. This is important because DHA-PC is the transport molecule for the DHA transport to the brain and the retina.

To explore the effects of enteral choline and DHA supplementation on plasma choline and DHA-PC concentrations, this randomized controlled study will assign 40 preterm infants to 1 of 4 groups: standard care, choline supplementation, DHA supplementation, and choline and DHA supplementation.

After 7 days of supplementation, a single dose of stable isotope labelled choline will be administered and the kinetics of newly synthesized DHA-PC determined to assess plasma levels, uptake and distribution of choline and DHA.

This study is designed to inform future larger studies evaluating this approach of enteral co-application of choline and DHA on important clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* preterm infants with a gestational age at birth between 24 and 32 weeks
* on almost complete enteral feeding (>75% of total fluid intake)

Exclusion Criteria:

* insufficient enteral intake,
* gastrointestinal disease,
* missing parental consent

Ages: 1 Week to 2 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
plasma concentrations of choline | following 7 days of supplementation

SECONDARY OUTCOMES:
de-novo DHA-phosphatidylcholine synthesis | following 7 days of supplementation at 12hours after D9-choline administration
DHA-phosphatidylcholine turnover | following 7.5 days of supplementation, from 12hours to 60 hours after D9-choline administration
fractions and concentrations of molecular species of phosphatidylcholine | baseline and following 7.5 and 10 days of supplementation
plasma concentrations of choline | baseline and following 7.5 and 10 days of supplementation
Plasma concentrations of betaine (a metabolite of choline) | baseline and following 7.5 and 10 days of supplementation
Plasma concentrations of dimethylglycine (a metabolite of choline) | baseline and following 7.5 and 10 days of supplementation
Plasma concentrations of trimethylamineoxide (TMAO, a metabolite of choline) | baseline and following 7.5 and 10 days of supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Axel Franz, MD, Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital of Tuebingen, Tübingen, Germany

REFERENCES:
- [Background] Bernhard W, Raith M, Kunze R, Koch V, Heni M, Maas C, Abele H, Poets CF, Franz AR. Choline concentrations are lower in postnatal plasma of preterm infants than in cord plasma. Eur J Nutr. 2015 Aug;54(5):733-41. doi: 10.1007/s00394-014-0751-7. Epub 2014 Aug 23. PMID 25148882
- [Background] Bernhard W, Raith M, Koch V, Kunze R, Maas C, Abele H, Poets CF, Franz AR. Plasma phospholipids indicate impaired fatty acid homeostasis in preterm infants. Eur J Nutr. 2014 Oct;53(7):1533-47. doi: 10.1007/s00394-014-0658-3. Epub 2014 Jan 24. PMID 24464176
- [Background] Bernhard W, Full A, Arand J, Maas C, Poets CF, Franz AR. Choline supply of preterm infants: assessment of dietary intake and pathophysiological considerations. Eur J Nutr. 2013 Apr;52(3):1269-78. doi: 10.1007/s00394-012-0438-x. Epub 2012 Sep 9. PMID 22961562
- [Derived] Bernhard W, Bockmann K, Maas C, Mathes M, Hovelmann J, Shunova A, Hund V, Schleicher E, Poets CF, Franz AR. Combined choline and DHA supplementation: a randomized controlled trial. Eur J Nutr. 2020 Mar;59(2):729-739. doi: 10.1007/s00394-019-01940-7. Epub 2019 Mar 11. PMID 30859363